CLINICAL TRIAL: NCT00177112
Title: Impact of Sterilization Technique on Incidence of Urinary Tract Infection After Cystoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Manoj Monga, MD, University of Minnesota
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0412M65852; 3519A
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-02-04 (Estimated); Status verified 2008-01

CONDITIONS: Urinary Tract Infections
Keywords: Cystoscopy
MeSH Terms: conditions — Urinary Tract Infections | interventions — Cystoscopy

INTERVENTIONS:
Procedure: clean patient preparation for cystoscopy
Procedure: sterile patient preparation for cystoscopy

SUMMARY:
The purpose of this study is to verify that the incidence rate of urinary tract infections after a routine outpatient cystoscopy is the same for non-sterile (clean) and sterile procedural techniques.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients undergoing routine outpatient flexible cystoscopy

Exclusion Criteria:

* Patients who have had a urinary tract infection within 3 months prior to flexible cystoscopy
* Patients with an indwelling catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2005-06; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To verify that the incidence rate of urinary tract infections after a routine outpatient cystoscopy is the same for non-sterile (clean) and sterile procedural techniques

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Anderson, MD, Principal Investigator — VAMC Minneapolis
Locations (1):
- VAMC Minneapolis, Minneapolis, Minnesota, United States